CLINICAL TRIAL: NCT02512705
Title: A Pilot Randomized Control Trial: The Ability to Medically Monitor With Use of Physical and Chemical Restraints or Seclusion of Acutely Agitated or Violent Patients Who Present to the Psychiatric Emergency Services
Brief Title: Medical Monitoring for Agitated Patients Pilot RCT - Medical Monitoring
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Janet Patterson, Medical Lead Psychiatric Emergency Services, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Patterson-1
Record Dates: First submitted 2015-07-23; First posted 2015-07-31 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Acute Agitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Seclusion Room (Other): The current practice is followed as a control group A.
  Interventions: Behavioral: Seclusion Room
- Physical Restraint (Experimental): Patient is placed in physical restraints to enable delivery of chemical restraints and medical monitoring and is monitored 1:1.
  Interventions: Device: Pinel Restraints

INTERVENTIONS:
Device: Pinel Restraints
  Arms: Physical Restraint
Behavioral: Seclusion Room
  Arms: Seclusion Room

SUMMARY:
The Psychiatric Emergency Services (PES) is an under researched area of clinical practice, largely in the management of acutely agitated and violent patients. The goal of this pilot randomized clinical trial (RCT) is to assess the benefit of medically monitoring patients that present with extreme agitation and/or violent behaviour to PES. Placing them in physical restraints and immediately administering chemical restraint, will enable medical monitoring of these potentially medically unstable patients. Investigators believe that this practice will provide safer management of patients, reduce risk to staff and other patients, reduce risk of undiagnosed medical conditions that underly the agitation, and increase clinical management and quality of care. Patients that come into the Emergency Department that are agitated and violent, where verbal-deescalation will not suffice, will be randomly treated with either immediate placement in seclusion (current practice) or be placed in physical restraints and given chemical restraint (as outlined in the BETA project guidelines). The same time interval assessments will be performed on both groups of patients including; medical monitoring and agitation scale assessment. Data will also be collected on number of violent episodes, code whites, required increase in the use of physical restraints, length of intervention, and more. This assessment will enable a comparison between the current practice and the proposed practice to establish evidence based clinical guidelines for the management of acute agitation in PES, where de-escalation techniques are ineffective and the lack of medical monitoring is harmful to the patient and can negatively effect their outcome. In order to best assess the importance of medical monitoring for such patients, a pilot study must be performed to assess the feasibility of such a phase III RCT study.

ELIGIBILITY:
Inclusion Criteria:

* Was agitated or violent upon entry into PES.
* Is 18+ years of age.
* Verbal de-escalation techniques are not useful for management of this patient.
* BETA Project techniques alone are not useful for management of this patient.
* The patient is assigned a CTAS1 or CTAS2 score.

Exclusion Criteria:

* The patient scores a "Low" or "Moderate" level of risk on the Violence/Aggression Screening Tool (VAST) that is used at ER triage.
* The point of agitation or violence began after the patient was already admitted to PES.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-09; Primary Completion 2015-12 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Analysis of feasibility, as measured by the recruitment rates | 3 months
  Process
Analysis of feasibility, as measured by staff and resource availability | 3 months
  Resources
Analysis of feasibility, as measured by baseline data of demographic and clinical characteristics | 3 months
  Scientific

SECONDARY OUTCOMES:
Occurrence of medical event | 3 months
  Were there any medical events? What was the time to the first medical event?
Time to medical event response | 3 months
  What was the time taken to respond to a medical event from the start of the intervention?
Time of agitation event response | 3 months
  What was the time it took to respond to an agitation event?